CLINICAL TRIAL: NCT02627729
Title: J-Pouch vs Side-to-End Anastomosis After Hand-Assisted Laparoscopic Low Anterior Resection for Rectal Cancer: Short and Long-Term Outcomes of a Prospective Randomized Trial
Brief Title: J-Pouch vs Side-to-End Anastomosis After Hand-Assisted Laparoscopic Low Anterior Resection for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nuri Okkabaz, MD, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DrLutfi2
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Quality of Life; Fecal Incontinence; Postoperative Complications
MeSH Terms: conditions — Fecal Incontinence; Postoperative Complications

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linear cutter-Circular stapler J pouch (Active Comparator): J pouch anal anastomosis after laparoscopic low anterior resection
  Interventions: Device: Linear cutter-Circular stapler
- Circular stapler Side-to-end anastomosis (Active Comparator): side to end coloanal anastomosis after laparoscopic low anterior resection
  Interventions: Device: Circular stapler

INTERVENTIONS:
Device: Linear cutter-Circular stapler — a 5 to 6 cm-long colonic pouch will be created with a 80 mm linear cutting-closing stapler. The anastomosis of j-pouch will be routinely strengthened with 3:0 vicryl sutures. Then, a pouch to anal anastomosis will be performed
  Arms: Linear cutter-Circular stapler J pouch
Device: Circular stapler — a 5 to 6 cm-long colonic segment will be left at the distal part and a side-to-end anastomosis will be performed.
  Arms: Circular stapler Side-to-end anastomosis

SUMMARY:
Current study aims to analyze the outcomes of j-pouch and side-to-end anastomosis in rectal cancer patients treated with laparoscopic hand-assisted low anterior resection

ELIGIBILITY:
Inclusion Criteria:

* patients with rectal cancer which is located up to 12 cm from the dentate line observed with a rigid rectosigmoidoscope

Exclusion Criteria:

* refusal of the patient to participate
* pregnancy,
* previous radiation therapy,
* those have cancers other than adenocarcinoma,
* those planned to have local excision or abdominoperineal resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-06; Primary Completion 2012-04 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Short Form 36 Quality of life Questionnaire | Change from baseline scores at 4th, 8th and 12th months after stoma reversal

SECONDARY OUTCOMES:
Postoperative complications | 30 days postoperatively
Functional outcome measured with Fecal Incontinence Severity Index | Change from baseline scores at 4th, 8th and 12th months after stoma reversal
Functional outcome measured with Sexual Health Inventory | Change from baseline scores at 4th, 8th and 12th months after stoma reversal
Functional outcome measured with Overactive Bladder validated 8 scale | Change from baseline scores at 4th, 8th and 12th months after stoma reversal